CLINICAL TRIAL: NCT07219238
Title: A Phase 2/3, Multicenter, Open-Label, Non-Randomized Study to Evaluate Diagnostic Performance of GEH300079 (68Ga) Injection Positron-Emission Tomography (PET)/Computed Tomography (CT) for Detection of Peritoneal Carcinomatosis (PC) in Patients With Colorectal, Gastric, Ovarian, or Pancreatic Cancers (PERISCOPE)
Brief Title: Study to Evaluate the Diagnostic Performance of GEH300079 (68Ga) Injection PET/CT for Detection of PC in Patients With Colorectal, Gastric, Ovarian, or Pancreatic Cancers (PERISCOPE)
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: Fortrea (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GE-282-201; IND:151901 (Other: US FDA); 2024-519384-18-00 (EU CTIS Number)
Record Dates: First submitted 2025-10-09; First posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Colorectal Cancer; Gastric Cancers; Ovarian Cancers; Pancreatic Ductal Adenocarcinoma
Keywords: Peritoneal Carcinomatosis (PC); Pancreatic Cancers; Colorectal cancer; Gastric cancer; FAPI; Ovarian cancer; 68Ga; PET/CT imaging; Diagnostic imaging; Diagnostic performance
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms; Ovarian Neoplasms; Peritoneal Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Masking Description: An independent, blinded read of the GEH300079 (68Ga) PET/CT and baseline SoC images will be performed at a central location (offsite) by independent readers blinded to the study information except the primary tumor site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GEH300079 (68Ga) PET/CT Injection (Experimental): Single IV bolus of GEH300079 (68Ga), target activity 3.6 MBq/kg (150-300 MBq). PET/CT scan at 60 ±5 min post-dose (vertex to mid-thigh, ~20-30 min). Phase 2 subset: additional scans at 15 ±5 min and 3 h ±10 min.
  Interventions: Drug: GEH300079 (68Ga) Injection Positron-Emission Tomography (PET)/Computed Tomography (CT)

INTERVENTIONS:
Drug: GEH300079 (68Ga) Injection Positron-Emission Tomography (PET)/Computed Tomography (CT) — Attenuation correction CT will commence after the administration of GEH300079 (68Ga), and immediately before the PET acquisition. The PET acquisition will encompass the participant's vertex through mid-thighs. Images will be acquired at 60 ±5 minutes post injection, with a scan duration of approximately 20 to 30 minutes.

SUMMARY:
This study is a Phase 2/3, prospective, multicenter, open-label, non-randomized clinical trial, in which GEH300079 (68Ga) PET/CT images will be acquired in patients with primary colorectal, gastric, ovarian, or Pancreatic Ductal Adenocarcinoma (PDAC) cancers and known or suspected Peritoneal Carcinomatosis (PC) before or after institutional Standard of Care (SoC) imaging. The primary objective is to evaluate the diagnostic performance of GEH300079 (68Ga) PET/CT for the detection of PC in patients with colorectal, gastric, or ovarian primary cancers, using a composite standard of truth (SoT), in a region-based analysis. The detection of PC in patients with primary PDAC will be explored in the Phase 2 part of the study.

The study is comprised of 2 distinct parts: Phase 2 aims to confirm the statistical and scientific assumptions for the Phase 3 part, and to confirm the optimal dose and timing of acquisition of GEH300079 (68Ga) PET/CT in the PC indication. Phase 2 includes 2 cohorts: Cohort A (participants with colorectal, ovarian and gastric primary cancer), and Cohort B (participants with primary PDAC), where analysis of Cohort B is descriptive only. Phase 3 aims to demonstrate the safety and efficacy of GEH300079 (68Ga) PET/CT for the detection of PC in patients with confirmed colorectal, gastric or ovarian primary cancers.

ELIGIBILITY:
Inclusion Criteria:

* Participant is ≥18 years of age
* Participant has provided signed informed consent before any study-specific screening procedures
* Participant has histopathologically confirmed primary colorectal, gastric or ovarian cancer or PDAC
* Participant has known or suspected PC from the tumor of origin. Suspicion may be based on imaging or clinical findings.
* Participant is scheduled for peritoneal surgery with curative intent, surgical exploration, or laparoscopy, with either: a. No neoadjuvant treatment received, treatment-naïve (i.e., undergoing upfront surgery or laparoscopy) b. Completed systemic treatment (which may include neoadjuvant chemotherapy) before GEH300079 ( 68Ga) PET/CT Imaging Visit
* Participant has Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Participant is able and willing to comply with all study procedures as described in the protocol

Exclusion Criteria:

* Participant is pregnant or breast-feeding, or sexually active and not using or not willing to use an acceptable form of birth control from screening up to 30 days after receiving the investigational medicinal product (IMP)
* Participant has a known disorder that, in the opinion of the investigator, will impact the study procedures
* Participant needs any intervention that would delay study participation
* Participant has non-resectable extra-abdominal metastasis and/or >3 hepatic metastases on standard work up
* Participant will not be able to complete the study, based on their anticipated life expectancy
* Participant has active bacterial, viral, or fungal infection requiring systemic antibacterial, anti-viral or antifungal therapy (topical medications are permitted)
* Participant has renal function impairment as defined by:

  1. For Phase 2: estimated glomerular filtration rate less than 60 mL/min
  2. For Phase 3: estimated glomerular filtration rate less than 30 mL/min
* Participant has severe hepatic function impairment as defined by:

  1. Aspartate aminotransferase (serum glutamic-oxaloacetic transaminase) and alanine aminotransferase (serum glutamic-pyruvic transaminase): ≤2.5 × upper limit of normal (ULN; ≤5 × ULN for participants with liver metastases)
  2. Bilirubin: ≤1.5 × ULN or direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN
* Participant has autoimmune disease that required systemic treatment in the past 2 years. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid) is allowed
* Participant has serious co-morbidities or serious non-malignant disease that in the opinion of the investigator, could compromise participant safety and/or protocol objectives
* Participant either received or is planning to receive any other investigational agent within the 28 days prior to the first imaging visit or during study participation (with the exception of the 3-month follow-up period)
* Participant has known or suspected hypersensitivity to any excipients used in GEH300079 (68Ga)
* Participant has severe claustrophobia, is unable to lie flat or fit into the scanner, or is unable to tolerate the PET/CT scan for any reason
* (Phase 3 only) Participant was previously included in Phase 2 of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Per-region sensitivity and Per-region specificity of GEH300079 (68Ga) PET/CT imaging to detect PC. | Single time point. Images will be acquired at 60 minutes ±5 minutes post injection, with a scan duration of approximately 20 to 30 minutes.
  The co-primary efficacy endpoint is based on region level sensitivity and specificity of GEH300079 (68Ga) PET/CT imaging for the detection of PC in participants with colorectal, gastric or ovarian primary cancer. GEH300079 (68Ga) PET/CT images collected during the Phase 2 part will be reviewed by 5 independent readers. Images collected during the Phase 3 part will be reviewed by 3 readers. The superiority of per region sensitivity (respectively specificity) to a pre-specified threshold of 75% (respectively 70%) will be assessed using one-sided Z-tests. The co-primary endpoints will be considered as met if superiority of both per region sensitivity and per region specificity is achieved by at least 3 of the 5 readers in the Phase 2 part, and by at least 2 of the 3 readers in the Phase 3 part.

SECONDARY OUTCOMES:
Superiority of the per region sensitivity of GEH300079 (68Ga) PET/CT to detect PC compared to baseline SoC imaging and non-inferiority of the per region specificity of GEH300079 (68Ga) PET/CT to detect PC compared to baseline SoC imaging. | Single time point. Baseline SoC images vs GEH300079 (68Ga) PET/CT Images acquired at 60 minutes ±5 minutes post injection, with a scan duration of approximately 20 to 30 minutes.
  Superiority of the per region sensitivity of GEH300079 (68Ga) PET/CT to detect PC compared to SoC imaging will be assessed on participants from the ITI using a McNemar test.
  Non-inferiority of the per region specificity of GEH300079 (68Ga) PET/CT to detect PC compared to SoC imaging, will be assessed using a restricted maximum likelihood estimate (RMLE) -based score test, with a non-inferiority margin of 10%.
  SoC images will be reviewed by 3 independent readers. The co-key secondary endpoints will be met if the co-primary endpoints are met and both co-key secondary endpoints are demonstrated for the same reader, for at least 2 of the 3 pairs of readers.
Superiority of the per participant sensitivity of GEH300079 (68Ga) PET/CT to detect PC compared to baseline SoC imaging in Phase 3 | Single time point. Baseline SoC images vs GEH300079 (68Ga) PET/CT Images acquired at 60 minutes ±5 minutes post injection, with a scan duration of approximately 20 to 30 minutes.
  Superiority of the per participant sensitivity of GEH300079 (68Ga) PET/CT to detect PC compared to baseline SoC imaging will be assessed using a McNemar test, in the Phase 3 part.
Per region PPV, NPV, and accuracy and per participant sensitivity, specificity PPV, NPV, and accuracy of GEH300079 (68Ga) PET/CT and baseline SoC imaging to detect PC | Single time point. Baseline SoC images vs GEH300079 (68Ga) PET/CT Images acquired at 60 minutes ±5 minutes post injection, with a scan duration of approximately 20 to 30 minutes.
  Per region PPV, NPV, and accuracy and per participant sensitivity, specificity PPV, NPV, and accuracy of GEH300079 (68Ga) PET/CT and baseline SoC imaging to detect PC will be tabulated.
Correlation between radiological and surgical/laparoscopic PCI scores | Single time point. Baseline SoC images. GEH300079 (68Ga) PET/CT Images acquired at 60 minutes ±5 minutes post injection, with a scan duration of approximately 20 to 30 minutes. Surgery/laparoscopy within 28 days post injection
  Correlation between radiological PCI scores (based on GEH300079 (68Ga) PET/CT, CT, MR, [18F]FDG PET/CT) and surgical/laparoscopic PCI score.
The number of Positive peritoneal regions and percentage of participants with a difference in the number of Positive peritoneal regions. | single time point. Baseline SoC images vs GEH300079 (68Ga) PET/CT Images acquired at 60 minutes ±5 minutes post injection, with a scan duration of approximately 20 to 30 minutes.
  The number of Positive peritoneal regions identified by GEH300079 (68Ga) PET/CT, CT, MR, and [18F]FDG PET/CT, and the percentage of participants with a difference in the number of Positive peritoneal regions identified by GEH300079 (68Ga) PET/CT and baseline SoC imaging.
SUVmax of GEH300079 (68Ga) PET/CT in comparison with [18F]FDG PET/CT. | Single time point Baseline [18F]FDG PET/CT images vs GEH300079 (68Ga) PET/CT Images acquired at 60 minutes ±5 minutes post injection, with a scan duration of approximately 20 to 30 minutes.
  SUVmax of GEH300079 (68Ga) PET/CT for the largest lesion identified within each peritoneal region from different primary cancers in comparison with [18F]FDG PET/CT.
SUVmean of GEH300079 (68Ga) PET/CT in comparison with [18F]FDG PET/CT. | Single time point Baseline [18F]FDG PET/CT images vs GEH300079 (68Ga) PET/CT Images acquired at 60 minutes ±5 minutes post injection, with a scan duration of approximately 20 to 30 minutes.
  SUVmean of GEH300079 (68Ga) PET/CT for the largest lesion identified within each peritoneal region from different primary cancers in comparison with [18F]FDG PET/CT.
SUVpeak of GEH300079 (68Ga) PET/CT in comparison with [18F]FDG PET/CT. | Single time point Baseline [18F]FDG PET/CT images vs GEH300079 (68Ga) PET/CT Images acquired at 60 minutes ±5 minutes post injection, with a scan duration of approximately 20 to 30 minutes.
  SUVpeak of GEH300079 (68Ga) PET/CT for the largest lesion identified within each peritoneal region from different primary cancers in comparison with [18F]FDG PET/CT.
Tumor to-background ratio (TBR) of GEH300079 (68Ga) PET/CT in comparison with [18F]FDG PET/CT. | Single time point Baseline [18F]FDG PET/CT images vs GEH300079 (68Ga) PET/CT Images acquired at 60 minutes ±5 minutes post injection, with a scan duration of approximately 20 to 30 minutes.
  TBR of GEH300079 (68Ga) PET/CT for the largest lesion identified within each peritoneal region from different primary cancers in comparison with [18F]FDG PET/CT.
Contrast-to-noise ratio (CNR) of GEH300079 (68Ga) PET/CT in comparison with [18F]FDG PET/CT. | Single time point Baseline [18F]FDG PET/CT images vs GEH300079 (68Ga) PET/CT Images acquired at 60 minutes ±5 minutes post injection, with a scan duration of approximately 20 to 30 minutes.
  CNR of GEH300079 (68Ga) PET/CT for the largest lesion identified within each peritoneal region from different primary cancers in comparison with [18F]FDG PET/CT.
Correlation between FAP expression and GEH300079 (68Ga) PET/CT uptake in PC from different primary cancer in Phase 2 | Single time point GEH300079 (68Ga) PET/CT Images acquired at 60 minutes ±5 minutes post injection, with a scan duration of approximately 20 to 30 minutes. Surgery/laparoscopy within 28 days post injection
  The correlation between GEH300079 (68Ga) PET/CT uptake in PC from different primary cancers and FAP expression measured by IHC in Phase 2.
Percentage of participants for whom GEH300079 (68Ga) PET/CT could have led to a change in treatment plan | Single time point GEH300079 (68Ga) PET/CT Images acquired at 60 minutes ±5 minutes post injection
Percentage of locoregional to systemic (M0 to M1) upstaging induced by GEH300079 (68Ga) PET/CT | Single time point GEH300079 (68Ga) PET/CT Images acquired at 60 minutes ±5 minutes post injection
GEH300079 (68Ga) PET/CT image quality at 15 ±5 minutes, 60 ±5 minutes, and 3 hour ±10 minutes post-injection, as well as for different simulated injected activities. | GEH300079 (68Ga) PET/CT Images acquired at 15 ±5 minutes, 60 ±5 minutes, and 3 hour ±10 minutes post-injection
  Visual assessment score of overall image quality at 15 ±5 minutes, 60 ±5 minutes, and 3 hours ±10 minutes post-injection, and across different simulated injected activities
Tumor to-background ratio (TBR) of GEH300079 (68Ga) PET/CT at 15 ±5 minutes, 60 ±5 minutes, and 3 hour ±10 minutes post-injection, as well as for different simulated injected activities | GEH300079 (68Ga) PET/CT Images acquired at 15 ±5 minutes, 60 ±5 minutes, and 3 hour ±10 minutes post-injection
  TBR for each GEH300079 (68Ga) PET/CT time point and each simulated injected activity
Contrast-to-noise ratio (CNR) of GEH300079 (68Ga) PET/CT TBR at 15 ±5 minutes, 60 ±5 minutes, and 3 hour ±10 minutes post-injection, as well as for different simulated injected activities. | GEH300079 (68Ga) PET/CT Images acquired at 15 ±5 minutes, 60 ±5 minutes, and 3 hour ±10 minutes post-injection
  CNR for each GEH300079 (68Ga) PET/CT time point and each simulated injected activity
Number of lesions detected by GEH300079 (68Ga) PET/CT at 15 ±5 minutes, 60 ±5 minutes, and 3 hour ±10 minutes post-injection, as well as for different simulated injected activities. | GEH300079 (68Ga) PET/CT Images acquired at 15 ±5 minutes, 60 ±5 minutes, and 3 hour ±10 minutes post-injection
  Count of lesions (<2 cm, ≥2 cm) for each GEH300079 (68Ga) PET/CT time point and each simulated injected activity
Size of lesions detected by GEH300079 (68Ga) PET/CT at 15 ±5 minutes, 60 ±5 minutes, and 3 hour ±10 minutes post-injection, as well as for different simulated injected activities. | GEH300079 (68Ga) PET/CT Images acquired at 15 ±5 minutes, 60 ±5 minutes, and 3 hour ±10 minutes post-injection
  Size of lesions for each GEH300079 (68Ga) PET/CT time point and each simulated injected activity
Coefficient of Variation (CV) of GEH300079 (68Ga) PET/CT SUV in Background and Reference Tissues at 15 ±5 minutes, 60 ±5 minutes, and 3 hour ±10 minutes post-injection, as well as for different simulated injected activities. | GEH300079 (68Ga) PET/CT Images acquired at 15 ±5 minutes, 60 ±5 minutes, and 3 hour ±10 minutes post-injection
  Variation coefficient of SUV in local background and reference tissues for each GEH300079 (68Ga) PET/CT time point and each simulated injected activity
Intra-reader reproducibility for GEH300079 (68Ga) PET/CT | Single time point GEH300079 (68Ga) PET/CT Images acquired at 60 minutes ±5 minutes post injection
  Cohen's kappa statistics with 95% CI for read vs re-read, for each of the readers.
Inter-reader agreement for GEH300079 (68Ga) PET/CT | Single time point GEH300079 (68Ga) PET/CT Images acquired at 60 minutes ±5 minutes post injection
  Cohen's kappa statistics with 95% CI for the assessment of agreement between 2 readers. Fleiss's kappa statistics with 95% CI will be provided for the assessment across the readers.

CONTACTS AND LOCATIONS:
Locations (2):
- BAMF Health, Grand Rapids, Michigan, United States
- Karolinska Universitetssjukhuset, Stockholm, Sweden